CLINICAL TRIAL: NCT06535815
Title: KetoNiFast: Impact of Cyclic Enteral Daytime Feeding With Ketogenic Nighttime Fasting on Outcome of Critical Ill Patients.
Brief Title: KetoNiFast: Cyclic Enteral Daytime Feeding With Ketogenic Nighttime Fasting
Acronym: KetoNiFast
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Sandra Emily Stoll, Dr., Assistant Professor, University Hospital of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-1398_1
Record Dates: First submitted 2024-07-23; First posted 2024-08-02 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Nutrition; Muscle Loss; Inflammatory Response
Keywords: Ketogenic diet; ketogenic fasting; cyclic enteral nutrition
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Intervention Model Description: Monocentric, prospective, randomized, interventional trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional: Cyclic enteral nutrition with ketogenic nighttime fasting (Active Comparator): Interventional group:
  12 hours of enteral feeding (as per patients´individual calorimetric requirements measured by indirect calorimetry) followed by a fasting period of 12 hours supported by the supplementation of exogenous ketone salts.
  Interventions: Other: Cyclic enteral feeding with nighttime fasting and exogenous ketone salt supplementation (ß-hydroxybutyrate)
- Control: Conventional continuous enteral nutrition (No Intervention): Control group Continuous enteral nutrition for 24 hours (as per patients´ individual caloric requirements defined by indirect calorimetry).

INTERVENTIONS:
Other: Cyclic enteral feeding with nighttime fasting and exogenous ketone salt supplementation (ß-hydroxybutyrate) — 12 hours of enteral feeding (as per patients´individual calorimetric requirements measured by indirect calorimetry) followed by a fasting period of 12 hours supported by the supplementation of exogenous ketone salts.
  Other Names: cyclic nutrition with nighttime fasting and exogenous ß-hydroxybutyrate supplementation
  Arms: Interventional: Cyclic enteral nutrition with ketogenic nighttime fasting

SUMMARY:
A physiological human nutrition includes circadian feeding and nighttime fasting during sleep. There is increasing evidence, that this natural fasting episode over nighttime majorly contributes to repair processes of the human body. So far, intensive care patients are normally enterally fed continuously, so that there is no circadian nutrition and no nighttime fasting. An enteral nutrition for 12 hours followed by a fasting period of 12 hours supported by exogenous ketone salts potentially improves the reconstitution of ICU patients compared to ICU patients who are continuously enterally fed.

DETAILED DESCRIPTION:
There is increasing evidence that a circadian rhythm of feeding (cyclic feeding) could be beneficial for critical ill patients. Cyclic feeding and fasting are assumed to have positive effects on the gut microbiome resulting in optimization of host responses to gastrointestinal pathogens. Another positive effect of cyclic feeding potentially results from activation of a "fasting response", inducing repair pathways such as ketogenesis, mitochondrial biogenesis, anti-inflammatory pathways, antioxidant defenses and autophagy processes. The activation of these repair pathways could diminish cellular stress and promote cellular recovery in critical ill patients. A randomized controlled trial by van Dyck et al. could show that fasting-mimicking intervals of 12 hours are sufficient to generate a metabolic fasting response without risking a caloric deficit. This fasting response can be enhanced by additional supplementation of exogenous ketones. A cyclic enteral nutrition with 12 hours of daytime feeding and 12 hours of ketogenic nighttime fasting compared to a continuous enteral feeding for 24 hours can potentially improve the reconstitution of critically ill Intensive Care patients. This improved reconstitution can be measured by maintenance of muscle mass (measured by ultrasound of the musculus rectus femoris), urea/creatinine ration, length of ventilation, length of ICU and hospital stay, 30-day mortality, ICU mobility scale.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent to participate in this study
* admission to ICU
* enteral nutrition

Exclusion Criteria:

* Severe liver dysfunction / liver failure (Child Pugh >7 points / category B)
* Severe kidney dysfunction (KDIGO stage 3)
* Total pancreatectomy / insulin dependent diabetes mellitus (IDDM)
* Pregnancy / lactation
* Hemoglobin concentration < 80g/l
* Severe metabolic disorders / severe autoimmune diseases
* Refractory metabolic or respiratory acidosis
* Dysfunction of mitochondrial transport of fatty acids
* Dysfunction of oxidation of fatty acids
* Dysfunction of gluconeogenesis, production and reduction of ketones
* Intermittent Porphyria
* Severe cardiac arrhythmias / cardiomyopathy
* Contraindication against enteral nutrition
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Loss of muscle mass | From date of randomization until the date of ICU discharge up to 1 month
  Loss of muscle mass via Ultrasound of M. rectus femoris of a predefined leg
Progress of urea / creatinine ratio | From date of randomization until the date of ICU discharge up to 1 month
  Urea / creatinine ratio in the patients´ blood

SECONDARY OUTCOMES:
Length of invasive and noninvasive ventilation | From date of randomization until the date of ICU discharge up to 1 month
  Length of invasive and noninvasive ventilation
Length of ICU and hospital stay | From date of randomization until the date of hospital discharge up to 6 months
  Length of ICU and hospital stay
30 day mortality on day 30 | From date of randomization 30 days
  30 day mortality on day 30
ICU mobility scale on discharge | From date of randomization until the date of ICU discharge up to 1 month
  ICU mobility scale (lowest score 0, highest score 10)

CONTACTS AND LOCATIONS:
Overall Officials: Bernd W Böttiger, Prof, Study Director — University Hospital Cologne
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No